CLINICAL TRIAL: NCT04240548
Title: Role of Regional Nodal Irradiation in Node Positive Breast Cancer Patients With ypN0 After Preoperative Chemotherapy
Brief Title: Radiation Therapy for ypN0 Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Rimoun Ramsis Anis Boutrus, Lecturer of Radiation Oncology, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-BC-1/2016
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; regional nodal irradiation; preoperative chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm: A (Experimental): regional nodal irradiation including axillary and supraclavicular lymph node groups along with chest wall or whole breast irradiation
  Interventions: Radiation: Regional Nodal Irradiation
- Arm: B (No Intervention): chest wall or whole breast only irradiation

INTERVENTIONS:
Radiation: Regional Nodal Irradiation
  Arms: Arm: A

SUMMARY:
This is a phase III randomized study comparing regional nodal irradiation vs. no irradiation for breast cancer patients presenting with node positive disease who turns into node negative after preoperative chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* WHO performance status 0-1
* Invasive Breast Cancer with cT1-3 cN1-2 at time of diagnosis
* Axillary nodal involvement can be detected using, clinical examination, ultrasound, CT scan or PET scan
* Pathologic confirmation using, FNAC, core biopsy or excisional biopsy
* ER, PR, Her2 neu and Ki67 status should be available for all patients
* All patients should have received standard preoperative chemotherapy prior to surgery
* At the time of surgery, all patients should have axillary clearance with at least 6 nodes harvested from the axilla
* Patients who have undergone mastectomy or lumpectomy with negative margins with ypN0, ypN0(+i) or ypN0(+mol) are eligible for randomization

Exclusion Criteria:

* Poor performance status
* Definitive clinical or radiologic evidence of metastatic disease
* T4 tumors including inflammatory breast cancer
* N3 disease detected clinically or by imaging
* Patients with histologically positive axillary nodes after preoperative chemotherapy
* Positive surgical margin after definitive surgery
* Previous ipsilateral or contralateral breast cancer
* Previous chest wall or breast irradiation
* Second primary cancer
* Active connective tissue disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Regional Nodal Failure ( axillary, internal mammary or supraclavicular recurrences ) | time from randomization till supraclavicular, axillary or internal mammary recurrence, assessed up to 10 years
  axillary, internal mammary or supraclavicular recurrences

SECONDARY OUTCOMES:
Disease Free survival | Time from randomization until local, regional or distant recurrence, assessed up to 10 years
  local recurrence, regional recurrence, distant recurrence, contralateral breast recurrence and second primary cancer
Overall Survival | from randomization till death from any cause, assessed up to 10 years
  death from any cause
Local Failure | from time of randomization until chest wall recurrence post mastectomy or In Breast Tumor Recurrence post lumpectomy, assessed up to 10 years
  chest wall recurrence post mastectomy or In Breast Tumor Recurrence post lumpectomy

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No